CLINICAL TRIAL: NCT07014436
Title: Prospective Cohort Study Evaluating Iron Supplementation in Patients With Altered Iron Status in the Context of Acute Inflammation (CARMI (CARence Martiale & Inflammation))
Acronym: CARMI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC25.0094
Record Dates: First submitted 2025-05-26; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Anemia; Inflammation
Keywords: cohort; anemia; inflammation; prospective; iron supplementation
MeSH Terms: conditions — Anemia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (iron supplementation): Patients who have received oral or IV iron as part of routine care for a ferritin between 30 and 300 µg/L and a transferrin saturation coefficient (TSC) < 20%.
- Group B (without iron supplementation): Patients who did not receive iron, despite a ferritin between 30 and 300 µg/L and a transferrin saturation coefficient (TSC) < 20%.

SUMMARY:
This study is a prospective, single center, open label cohort study evaluating iron supplementation in patients with impaired martial status in the acute inflammatory setting.

The main objective of this study is to evaluate the effectiveness of iron supplementation in anemic patients with inflammation and an altered iron status in the 'grey zone,' defined by a ferritin level between 30 and 300 µg/L and a transferrin saturation coefficient (TSC) of less than 20%, in the patient internal medicine/general medicine unit of the Grenoble Alpes University Hospital.

The primary endpoint is the difference in hemoglobin levels at 3 months after hospital discharge between patients treated with or without martial supplementation.

We hypothesize that iron supplementation more effectively improves hemoglobin levels at three months compared to no supplementation in patients with anemia and altered iron status (ferritin between 30 and 300 µg/L and a transferrin saturation coefficient (TSC) < 20%) in the context of acute inflammation.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the effectiveness of iron supplementation in anaemic patients with inflammation and an altered iron status.

The primary endpoint is the difference in hemoglobin levels at 3 months after hospital discharge between patients treated with or without martial supplementation, and our hypothesis is that iron supplementation improves hemoglobin levels at three months compared to no supplementation in patients with anaemia and altered iron status (ferritin between 30 and 300 µg/L and a transferrin saturation coefficient (TSC) < 20%) in the context of acute inflammation.

The secondary objectives are to evaluate the effectiveness of iron supplementation in anaemic and inflammatory patients with iron status in the "grey zone" (ferritin between 30 and 300 µg/L and a transferrin saturation coefficient (TSC) < 20%), to identify demographic, clinical, and biological factors associated with the correction of anaemia in the iron-treated group, to identify demographic, clinical, and biological factors associated with the correction of anaemia in the non-iron-treated group and to assess the safety of iron supplementation.

Anemic patients (hemoglobin < 13 g/dL in men and < 12 g/dL in women), with inflammation (CRP > 30 mg/L), and iron status in the "grey zone" (ferritin between 30 and 300 µg/L and transferrin saturation < 20%) within the first three days of hospitalization are observed according to the iron supplementation strategy chosen as part of their routine care, allowing for a retrospective classification into two groups:

* Group A: patients who received iron supplementation despite having ferritin between 30 and 300 µg/L and transferrin saturation coefficient (TSC) < 20%.
* Group B: patients who did not receive iron supplementation despite ferritin between 30 and 300 µg/L and transferrin saturation coefficient (TSC) < 20%.

Sociodemographic and clinical data of the patients in each group will be collected to control for potential confounding factors in the statistical analysis.

Patients are included the day before or at the end of their hospital stay, once all medical decisions-including whether or not to administer iron-have been made independently of the study. No influence is exerted on therapeutic choices, which are based solely on the routine practices of hospital physicians.

ELIGIBILITY:
Inclusion Criteria :

* Anemia (Hb < 130 g/L in men and < 120 g/L in women) within the first 3 days of hospitalization in the department
* Biological signs of inflammation (CRP ≥ 30 mg/L) within the first 3 days of hospitalization in the department
* Ferritin between 30 and 300 µg/L and a transferrin saturation coefficient (TSC) < 20% within the first 3 days of hospitalization in the department

Exclusion Criteria :

* Patients who object to the use of their data for research purposes
* Patients unable to provide informed consent to participate in the research
* Patients who received a red blood cell transfusion during hospitalization or in the month prior
* Patients receiving erythropoietin (EPO) treatment
* Patients treated with iron supplementation within one month prior to hospitalization
* Congenital hemoglobinopathy (e.g., thalassemia, sickle cell disease)
* Chemotherapy within the past 3 months or planned chemotherapy within the next 3 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included in the study will be recruited from patients hospitalised in the various units of the Internal and Polyvalent Medicine Department at Grenoble Alpes University Hospital (Internal Medicine 3eA, Post-Emergency Unit 3eB and Internal Medicine 3eC).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean increase in hemoglobin | At 3 months (end of study)
  The improvement in anemia, represented by the mean hemoglobin level (g/L) measured at 3 months after hospitalization, between patients who received iron supplementation and those who did not.
  * Analysis population : All included patients
  * Statistical tests:
  * Student's t-test if the data are normally distributed with homogeneity of variances, particularly for hemoglobin.
  * Wilcoxon non-parametric test if normality assumptions are not met.
  * Multivariate analysis (ANCOVA) adjusted for potential confounding factors (age, sex, comorbidities, baseline CRP, baseline ferritin, baseline transferrin saturation coefficient (TSC)).

SECONDARY OUTCOMES:
Correction of anemia : | At 3 months (end of study)
  Proportion of patients having corrected their anemia (hemoglobin level ≥ 13 g/dL in men, ≥ 12 g/dL in women).
  * Population : All included patients
  * Test : Comparison of proportions (Chi-squared test or Fisher's exact test, depending on whether normality assumptions are met
Identify factors associated with anemia correction | At 3 months (end of study)
  Analysis of demographic (age, gender), clinical (comorbidities) and biological factors
  * Population : Treated and untreated subgroups
  * Test : Exploratory analysis using logistic regression
Adverse events : | At 3 months (end of study)
  Incidence of adverse effects associated with iron supplementation (hypersensitivity, iron overload).
  * Population : Treated patients
  * Test : Descriptive analysis (counts, percentages)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis BOCQUET, Hospital Doctor, Principal Investigator — University Hospital, Grenoble Alpes
Locations (1):
- University Hospital, Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fletcher A, Forbes A, Svenson N, Wayne Thomas D; A British Society for Haematology Good Practice Paper. Guideline for the laboratory diagnosis of iron deficiency in adults (excluding pregnancy) and children. Br J Haematol. 2022 Feb;196(3):523-529. doi: 10.1111/bjh.17900. Epub 2021 Oct 24. No abstract available. PMID 34693519
- [Background] Kiani AK, Dhuli K, Donato K, Aquilanti B, Velluti V, Matera G, Iaconelli A, Connelly ST, Bellinato F, Gisondi P, Bertelli M. Main nutritional deficiencies. J Prev Med Hyg. 2022 Oct 17;63(2 Suppl 3):E93-E101. doi: 10.15167/2421-4248/jpmh2022.63.2S3.2752. eCollection 2022 Jun. PMID 36479498
- [Result] Shepshelovich D, Rozen-Zvi B, Avni T, Gafter U, Gafter-Gvili A. Intravenous Versus Oral Iron Supplementation for the Treatment of Anemia in CKD: An Updated Systematic Review and Meta-analysis. Am J Kidney Dis. 2016 Nov;68(5):677-690. doi: 10.1053/j.ajkd.2016.04.018. Epub 2016 Jun 16. PMID 27321965
- [Result] Romanet T, Bedouch P, Zaoui P. [Assessment of iron deficiency anemia management in the general hospital of Grenoble: A 12-month follow-up of an intravenous ferric carboxymaltose treatment program in a cohort of patients with non-dialysis-dependent chronic kidney disease]. Nephrol Ther. 2019 Apr;15(2):104-109. doi: 10.1016/j.nephro.2018.10.006. Epub 2019 Feb 23. French. PMID 30803900
- [Result] Agrawal S, Sonawane S, Kumar S, Acharya S, Gaidhane SA, Wanjari A, Kabra R, Phate N, Ahuja A. Efficacy of Oral Versus Injectable Iron in Patients With Chronic Kidney Disease: A Two-Year Cross-Sectional Study Conducted at a Rural Teaching Hospital. Cureus. 2022 Jul 31;14(7):e27529. doi: 10.7759/cureus.27529. eCollection 2022 Jul. PMID 36060352
- [Result] Sieske L, Janssen G, Babel N, Westhoff TH, Wirth R, Pourhassan M. Inflammation, Appetite and Food Intake in Older Hospitalized Patients. Nutrients. 2019 Aug 22;11(9):1986. doi: 10.3390/nu11091986. PMID 31443557
- [Result] Petry N, Olofin I, Hurrell RF, Boy E, Wirth JP, Moursi M, Donahue Angel M, Rohner F. The Proportion of Anemia Associated with Iron Deficiency in Low, Medium, and High Human Development Index Countries: A Systematic Analysis of National Surveys. Nutrients. 2016 Nov 2;8(11):693. doi: 10.3390/nu8110693. PMID 27827838
- See also: " HAS 2011 - Choix des examens du métabolisme du fer en cas de suspicion de carence martiale - texte long ", s. d. — https://www.has-sante.fr/upload/docs/application/pdf/2011-11/texte_court__bilan_martial_carence_2011-11-09_17-22-2_135.pdf
- See also: KIANI et al., " Main nutritional deficiencies ". — https://pubmed.ncbi.nlm.nih.gov/36479498/
- See also: " Revue Médicale Suisse 2011 ; 7 : 2018-23 RMS_idPAS_D_ISBN_pu2011-37s_sa03_art03.pdf " — https://www.revmed.ch/view/514249/4206039/RMS_idPAS_D_ISBN_pu2011-37s_sa03_art03.pdf
- See also: " HAS 2011 - Choix des examens du métabolisme du fer en cas de suspicion de carence martiale - texte long " — https://www.has-sante.fr/upload/docs/application/pdf/2011-11/texte_court__bilan_martial_carence_2011-11-09_17-22-2_135.pdf
- See also: World Health Organization, WHO Guideline on Use of Ferritin Concentrations to Assess Iron Status in Individuals and Populations (Geneva: World Health Organization, 2020) — https://iris.who.int/handle/10665/331505
- See also: Aurelien Amiot et al., " Practice guidelines for the diagnosis and management of ulcerative colitis " 29 (2022). — https://www.researchgate.net/publication/363319366_Practice_guidelines_for_version_longue_the_diagnosis_and_management_of_ulcerative_colitis
- See also: " KDIGO-2012-Anemia-Guideline-English.pdf ", consulté le 24 novembre 2024 — https://kdigo.org/wp-content/uploads/2016/10/KDIGO-2012-Anemia-Guideline-English.pdf
- See also: " 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure | Journal de Cardiologie " — https://pubmed.ncbi.nlm.nih.gov/34447992/
- See also: "ANSM 1997 - Hémogramme " — https://www.has-sante.fr/upload/docs/application/pdf/Hemogram.pdf